CLINICAL TRIAL: NCT01054001
Title: Early Start of Oral Sildenafil 100mg for Erectile Dysfunction After Robotic Assisted Laparoscopic Radical Prostatectomy
Acronym: SILRALP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Sang Eun Lee, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WS486539
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostatectomy; erectile dysfunction
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early (Active Comparator): men with on- demand sildenafil 100mg dosing from the early postoperative period
  Interventions: Drug: sildenafil 100mg
- Delayed (Active Comparator): men with on- demand sildenafil 100mg dosing from the delayed postoperative period
  Interventions: Drug: sildenafil 100mg

INTERVENTIONS:
Drug: sildenafil 100mg — sildenafil 100mg per oral twice a week
  Other Names: Viagra 100mg

SUMMARY:
The investigators try to investigate the benefit of early administration (immediately after urethral catheter removal) of sildenafil after nerve-sparing RALP for 3 months. The investigators will compare the potency rates up to 2 years after nerve-sparing RALP in men with on- demand sildenafil 100mg dosing from the early postoperative period (immediately after urethral catheter removal) with from the delayed postoperative period (3 months after RP).

DETAILED DESCRIPTION:
Various studies using animal models of CN neuroparaxia and clinical trials have demonstrated somewhat beneficial effect of PDE-5 inhibitors on smooth muscle cells of the corpus cavernosum. PDE-5 inhibitors including sildenafil have demonstrated the effectiveness in the management of postprostatectomy ED. In the animal experiments, PDE-5 inhibitors lowered the severity of the fibrosis in the corpus cavernosum of rats with CN cutting. In the clinical trials, on-demand dosing or routine dosing of PDE-5 inhibitors improved the potency rates in men received NSRP, and improvements of the potency rate did not appear to be statistically different among two dosing regimens.

But, there are few studies on the potency rate according to the start time of the administration of PDE-5 inhibitors (eg. early vs. delayed post-operative dosing). At present, it is not conclusive that whether nerve-sparing RALP provides more higher potency rate than conventional surgery in men with prostate cancers. But, with more precise dissection of CN, the robotic surgery appears to have more chances to maintain the potency in men received RP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with agree to participate with the study
* Korean male subjects aged 50 years or older with clinically localized prostate cancer
* Preoperative potent men (IIEF-5 score 17 or more than 17)
* Patients in a stable, heterosexual relationship with a single partner for at least the past six months
* Suitable for nerve sparing indication

Exclusion Criteria:

* Genital anatomical deformities that would significantly impair erection
* Other sexual disorders (e.g. hypoactive sexual desire) that are considered to be the primary diagnosis when there is a coexisting diagnosis of erectile dysfunction.
* Known raised prolactin level (>3 times the upper limit of the normal range) or low free testosterone level (confirmed to be >20% below the lower limit of the normal range on blood collected between 09:00 and 11:00 hours).
* Major psychiatric disorder (including major depression or schizophrenia) that is not well controlled on treatment.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
patterns of recovery of erectile functions after nerve sparing RALP in men with on- demand sildenafil 100mg dosing from the early postoperative period (using IIEF-5) | 1 year

SECONDARY OUTCOMES:
comparison of the potency rates in men with on- demand sildenafil 100mg dosing from the early postoperative period with from the delayed postoperative period | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Sang Eun Lee, Professor, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyeonggido, South Korea